CLINICAL TRIAL: NCT06429553
Title: A Multicenter Randomized Controlled Clinical Study of Minimally Invasive Intracranial Hematoma Aspiration and Drainage Combined With Urokinase Injection and Drug Therapy for Spontaneous Intracerebral Hemorrhage
Brief Title: Minimally Invasive Intracranial Hematoma Aspiration for Spontaneous Intracerebral Hemorrhage
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023KY135
Record Dates: First submitted 2024-05-05; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Spontaneous Cerebral Hemorrhage
Keywords: Spontaneous cerebral hemorrhage; intracranial hematoma aspiration; urokinase
MeSH Terms: interventions — Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hematoma puncture group (Experimental): Minimally invasive hematoma aspiration drainage combined with urokinase injection
  Interventions: Procedure: Minimally invasive hematoma aspiration drainage combined with urokinase injection
- Drug conserved group (Sham Comparator): Drug conserved group
  Interventions: Procedure: Minimally invasive hematoma aspiration drainage combined with urokinase injection

INTERVENTIONS:
Procedure: Minimally invasive hematoma aspiration drainage combined with urokinase injection — Minimally invasive hematoma aspiration drainage combined with urokinase injection

SUMMARY:
To observe the effect of minimally invasive intracranial hematoma aspiration and drainage combined with urokinase injection and drug therapy on prognosis of spontaneous cerebral hemorrhage.

DETAILED DESCRIPTION:
Intracerebral hemorrhage (ICH) refers to the spontaneous rupture of large and small arteries, veins, and capillaries in the brain caused by various reasons under non-traumatic conditions. Hypertension is the most common predisposing factor for intracerebral hematoma, and the risk increases with age. The challenge in surgical hematoma evacuation lies in the potential for surgical complications to negate the benefits of hematoma removal. Surgical treatment is generally considered only when the supratentorial hematoma causes a life-threatening space-occupying effect. Therefore, the size of the intracerebral hematoma is a key factor in determining whether surgery can bring benefits to patients. Specifically, intracerebral hematomas with a volume less than 30 ml are considered small and medium-sized.

Previously, drug-based conservative treatment was often the first choice for small and medium-sized intracerebral hematomas. However, with the accumulation of clinical data, it has been found that while these patients have low blood loss and mortality, their neurological function impairment is significant, and the recovery of neurological function under conservative treatment is often suboptimal. Therefore, some scholars have suggested the use of adjunctive surgical options for small and medium-sized intracerebral hematomas, such as small craniotomy, craniotomy, endoscopic surgery, fibrinolytic therapy combined with hematoma aspiration, and CT-guided stereotactic aspiration (i.e., minimally invasive surgery).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 years;
2. ICH in the basal ganglia was diagnosed by CT examination of the head (bleeding mainly from the caudate nucleus, lentiform nucleus, clavate nucleus or amygdala);
3. Based on CT examination of the head, the volume of hematoma was calculated to be 20-40 mL, and the midline structure was shifted horizontally in the pineal gland < 3 mm; The calculation formula of hematoma volume V (cm3) = A*B*C*1/2, where A is the longest diameter (cm) of the largest level of hematoma in the horizontal CT scan, B is the widest diameter (cm) of the hematoma in the plane perpendicular to A, and C is the thickness (cm) of the hematoma in the CT film;
4. The time from onset to randomization is within 48 hours;
5. GCS score 4-14 points during randomization;
6. NIHSS score >= 6 points during randomization;
7. Muscle strength of unilateral limbs on the symptomatic side is grade 0-3;
8. mRS0-1 score before onset;
9. Systolic blood pressure was controlled below 180mmHg before randomization;
10. Written informed consent signed by the patient and his legal representative.

Exclusion Criteria:

1. Bleeding in other areas (such as the thalamus, brain stem, or cerebellum);
2. Bleeding caused by other causes (such as aneurysm, arteriovenous malformation, brain trauma, brain tumor, hemorrhage transformation of massive cerebral infarction, hemorrhage caused by amyloidosis, hemorrhage caused by coagulation disorder) or combined with aneurysm, arteriovenous malformation, brain trauma, brain tumor, massive cerebral infarction, amyloidosis, severe coagulation disorder;
3. Recent history of cerebral hemorrhage (< 1 year);
4. Multiple intracranial hemorrhage;
5. The CTA source map indicated early signs of expanded intracerebral hemorrhage hematoma (point sign), and the possibility of progressive hemorrhage was largely ruled out;
6. Patients with ventricular hemorrhage or ICH intrusion into the ventricle should be considered for external ventricular drainage;
7. Any history of parenchyma or other intracranial subarachnoid, subdural or epidural blood and surgical history within the last 30 days;
8. Patients with coagulation dysfunction such as hereditary or acquired bleeding constitution and lack of coagulation factor;
9. Hemoglobin < 100 g/L, hematocrit < 25%, platelet count < 100*10^9/L;
10. Were receiving anticoagulant drugs such as warfarin, dabigatran or rivaroxaban within one week before enrollment, with INR > 1.4;
11. Long-term anticoagulant and antiplatelet therapy is expected;
12. There is a history of internal bleeding, such as digestive tract bleeding, urogenital system bleeding, respiratory tract bleeding is not completely controlled;
13. Myocardial infarction within the last 30 days;
14. Known high risk of embolism, including patients with mechanical heart valve implantation, history of left heart thrombosis, mitral stenosis with atrial fibrillation, acute pericarditis, or subacute bacterial endocarditis. Atrial fibrillation without mitral stenosis is suitable;
15. Severe liver function damage, ALT > 3 times the upper limit of normal, or AST > 3 times the upper limit of normal. Severe renal insufficiency, glomerular filtration rate < 30 ml/min/1.73m2;
16. Hypertension that could not be effectively controlled by active antihypertensive therapy before randomization (systolic blood pressure was still greater than 180 mmHg);
17. Patients with Alzheimer's disease or mental illness are unable to complete the follow-up plan as required;
18. Combined with any serious diseases that may be assessed to interfere with the test results: including diseases of the respiratory system, circulatory system, digestive system, genitourinary system, endocrine system, immune system and blood system;
19. Those who currently have drug or alcohol abuse or dependence and are expected to have poor compliance and difficulty in completing follow-up;
20. Allergic to urokinase or surgery-related drugs and instruments;
21. Pregnant or lactating women, or those planning to become pregnant within one year;
22. Life expectancy of < 12 months due to advanced stage of any disease;
23. Are participating in other clinical trials or have been included in this trial in the previous stage;
24. The patient or his legal guardian is not willing to sign a written informed consent (YNMT).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale score (mRS)（0-6）（ higher scores mean a worse outcome.） | 6 months
  Modified Rankin Scale score (mRS)（0-6）（ higher scores mean a worse outcome.）

SECONDARY OUTCOMES:
volume of hematoma | 2 weeks
  volume of hematoma
National Institutes of Health Stroke Scale（NIHSS)（0-42）（ higher scores mean a better outcome.） | 6 months
  National Institutes of Health Stroke Scale（NIHSS)（0-42）（ higher scores mean a better outcome.）
Muscle strength classification change（0-5）（ higher scores mean a better outcome.） | 6 months
  Muscle strength classification change（0-5）（ higher scores mean a better outcome.）

CONTACTS AND LOCATIONS:
Locations (1):
- Hao Xu, Hefei, Anhui, China